CLINICAL TRIAL: NCT03938012
Title: Evaluating Mutations in MET and TP53 Among Patients Diagnosed With Squamous Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/00640
Record Dates: First submitted 2019-04-05; First posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Squamous Cell Carcinoma of the Lung; Squamous Cell Carcinoma of the Head and Neck
Keywords: mutations in MET and TP53
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patient blood was also required for extraction of cell free DNA (cfDNA) and genomic DNA (gDNA).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung and head and neck tumours: 1. Age 18 years or older
  2. Histologic or cytologic confirmation of metastatic squamous cell carcinoma of the lung or head and neck region
  3. No other active malignancy within the past 24 months
  4. Refractory disease

SUMMARY:
This study focuses on advanced lung and head and neck SCC tumours, with adjacent normal lung tissues. Biopsies will be performed in National University Health System, Singapore (NUHS) as part of participants' standard care. Patient blood was also required for extraction of cell free DNA (cfDNA) and genomic DNA (gDNA). Patients' medical records will also be reviewed for the purpose of this study.

DETAILED DESCRIPTION:
Primary objective:

To investigate the prevalence of MET and TP53 mutations, as well as HER2 and MET amplification, in lung and head and neck tumours, through prospective collection of tumour specimens in newly recruited patients.

Secondary objectives:

1. To distinguish the presence of somatic/germline MET and TP53 mutation in lung and head and neck tumours.
2. To detect for amplifications of MET and/or HER2 genes in SCC samples.
3. To investigate the association and interaction of cMet and HER2 in SCC tumours.
4. To establish a prospective documation of clinical, histopathological, treatment and follow-up (clinic pathological) data of newly recruited patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Histologic or cytologic confirmation of metastatic squamous cell carcinoma of the lung or head and neck region
3. No other active malignancy within the past 24 months
4. Refractory disease

Exclusion Criteria:

1. Patient with other active malignancy within the past 24 months
2. Unable or unwilling to provide signed informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study intend to recruit a total of 80 patients over 2 years. Written informed consent will be requested from every patient prior to enrollment into the study. All eligibility criteria and consent form must be met before tumour DNA and plasma DNA from patients can be processed.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-10-03 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Identification of MET mutation using digital droplet PCR (ddPCR) | 2 years
  Germline DNA from the patients will be harvested from whole blood, and the polymorphic MET variant will be determined using ddPCR. Customised probes detecting wildtype MET allele or MET-N375S allele are designed to for genotyping (homozygous/heterozygous).
Identification of TP53 mutation using Sanger sequencing | 2 years
  DNA from the tumour specimens will be harvested for sequencing to identify cases with somatic mutations of TP53 gene. Changes in codon sequences will be reported.
Presence of MET and HER2 amplification using fluorescence in situ hybridization (FISH) | 2 years
  FFPE samples retrieved from patients genotyped with MET-N375S polymorphism will be subjected to MET and HER2 testing Abbott PathVysion DNA test kits. Data will be analysed with fluorescence microscopy. HER2 amplification will be defined as gene copies versus chromosome 17 polysomy. MET amplification will be defined as gene copies per nucleus.
Interaction of MET and HER2 receptor tyrosine kinases using proximity ligation assay (PLA) | 2 years
  PLA will be performed using DUOLINK in situ hybridization. Validation MET and HER2 antibodies will be used for the assay, and signal will be detected with fluorescence microscopy. Detection and quantification of positive signals will determine the presence of MET-HER2 interaction in clinical specimens.
Cell free DNA (cfDNA) will be extracted from patients' plasma to detect for presence of somatic/germline mutation | 2 years
  Extracted cfDNA will be subjected to ddPCR using designed probes for MET and TP53 mutations. Copies of cfDNA/1mL of plasma will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Boon Cher Goh, Principal Investigator — Study Principal Investigator
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stransky N, Egloff AM, Tward AD, Kostic AD, Cibulskis K, Sivachenko A, Kryukov GV, Lawrence MS, Sougnez C, McKenna A, Shefler E, Ramos AH, Stojanov P, Carter SL, Voet D, Cortes ML, Auclair D, Berger MF, Saksena G, Guiducci C, Onofrio RC, Parkin M, Romkes M, Weissfeld JL, Seethala RR, Wang L, Rangel-Escareno C, Fernandez-Lopez JC, Hidalgo-Miranda A, Melendez-Zajgla J, Winckler W, Ardlie K, Gabriel SB, Meyerson M, Lander ES, Getz G, Golub TR, Garraway LA, Grandis JR. The mutational landscape of head and neck squamous cell carcinoma. Science. 2011 Aug 26;333(6046):1157-60. doi: 10.1126/science.1208130. Epub 2011 Jul 28. PMID 21798893
- [Result] Cancer Genome Atlas Research Network. Comprehensive genomic characterization of squamous cell lung cancers. Nature. 2012 Sep 27;489(7417):519-25. doi: 10.1038/nature11404. Epub 2012 Sep 9. PMID 22960745